CLINICAL TRIAL: NCT04225351
Title: Treatment of Multiple Gingival Recession Defects With a Coronally Advanced Flap or a Modified Tunnel Technique and a Volume Stable Three-dimensional Xenogeneic Collagen Matrix: a Monocentric Randomized Clinical Trial
Brief Title: Treatment of Multiple Gingival Recessions With a MCAF or a MCAT and a Collagen Matrix
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo de Sanctis, Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fibro-gide 1
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCAF+CM (Experimental): Modified coronally advanced flap + collagen matrix
  Interventions: Procedure: MCAF+CM
- MCAT+CM (Active Comparator): Modified coronally advanced tunnel technique + collagen matrix
  Interventions: Procedure: MCAT+CM

INTERVENTIONS:
Procedure: MCAF+CM — CAF procedure + collagen matrix
  Arms: MCAF+CM
Procedure: MCAT+CM — Tunnel procedure + collagen matrix
  Arms: MCAT+CM

SUMMARY:
In a recent meta-analysis, Graziani et al. reported that despite the "ideal" treatment for multiple gingival recession defects is not yet identified, there are some indirect suggestions from the analyzed data that, in comparison to the traditional coronally advanced flap (CAF) approach, the use of additional grafting, modifications of the flap technique or tunnel variation with connective tissue graft (CTG) may improve clinical results.

Furthermore, various allografts or replacement biomaterials have been developed instead of a connective tissue graft in order to reduce patient morbidity. A newly developed porcine-derived bio-resorbable collagen matrix (CM) (Fibro-Gide) has been recently introduced as an alternative to CTG in periodontal plastic surgery.

The aim of this study will be to compare the outcomes of two muco-gingival surgery techniques, the modified coronali advanced flap (MCAF) for multiple recession defects and the modified coronally advanced tunnel technique (MCAT), performed in the Department of Periodontology of San Raffaele Hospital with the results reported in the literature.

Secondarily, the study will evaluate whether patients report a preference in terms of discomfort and perception of aesthetics between the two surgical techniques.

DETAILED DESCRIPTION:
The present research is a monocentric prospective parallel randomized controlled clinical trial.

Patients presenting multiple gingival recessions in the maxillary will be enrolled in the study after having signed an informed consent. Recessions will be treated by means of two mucogingival surgery techniques: modified coronally advanced flap (MCAF) and modified coronally advanced tunnel technique (MCAT), in association with the use of a collagen matrix (CM).

Two experienced practitioners (M.d.S. and S.A.) will perform the surgical session according to the technique as presented by Zucchelli & de Sanctis 2000 and Aroca et al. 2013.

- Modified coronally advanced flap (MCAF): After local anesthesia, a horizontal incision is made to include one tooth on each side of the teeth to be treated. The horizontal incision of the envelope flap consists of oblique sub-marginal incisions in the interdental areas, incisions which continue with the intra-sulcular incision at the recession defects.

Each surgical papilla (SP) is dislocated with respect to the anatomic papilla by the oblique sub-marginal interdental incisions; in particular, the surgical papilla mesial to the flap midline are dislocated more apically and distally, while the papilla distal to the mid-line are shifted in a more apical and mesial position.

The envelope flap is raised with a split-full-split approach in the coronal-apical direction: the surgical papilla is dissected in a split-thickness manner, while gingival tissue apical to the root exposures is raised in a full-thickness manner (to provide that portion of the flap critical for root coverage with more thickness). Finally, the most apical portion of the flap is elevated in a split-thickness manner to facilitate the coronal displacement of the flap.

The portion of the root exposure with loss of clinical attachment (gingival recession plus probeable gingival sulcus/pocket) are mechanically treated with the use of curettes and EDTA is applied for 2 minutes.

The remaining tissue of the anatomic interdental papilla is de-epithelialized to create connective tissue beds to which the surgical papilla are sutured.

A sharp dissection into the vestibular lining mucosa is then carried out to eliminate muscle tension. Flap mobilization is considered "adequate" when the marginal portion of the flap is able to passively reach a level coronal to the cemento-enamel junction (CEJ) at each single tooth in the surgical site. The flap, in fact, should be stable in its final position even without the sutures.

The porcine-derived bio-resorbable collagen matrix (CM) (Fibro-Gide) is now prepared for placement on the interested areas: the width of the matrix must be reduced to 3-4 mm and the matrix has to adapt to the receiving tissues, when placed, a suture (6/00) must be used to hold it in position.

Sling sutures (6/00) are performed to accomplish a precise adaptation of the buccal flap on the exposed root surfaces and to stabilize every single surgical papilla over the interdental connective tissue bed.

- Modified coronally advanced tunnel technique (MCAT): Immediately before surgery, composite stops are placed at the contact points to prevent collapse of the future suspended sutures into the inter-proximal spaces.

After local anaesthesia, root planing of the exposed root surface is performed by means of hand instruments. Ethylenediaminetetraacetic (EDTA) is applied on the sites.

Subsequently, intra-sulcular incisions were placed and muco-periosteal flap separation are raised using sharp tunnel elevators. The muco-periosteal dissection is extended beyond the muco-gingival junction (MGJ) and under each papilla, to allow passive, tension-free mobilization in coronal direction. Muscle fibres and any remaining collagen bundles on the inner aspect of the flap alveolar mucosa are cut using Gracey curettes with extreme care in order to obtain a passive coronal positioning of the flap and the papilla and to avoid perforation of the flap.

The porcine-derived bio-resorbable collagen matrix (Fibro-Gide) is now prepared for placement on the interested areas: the width of the matrix must be reduced to 3-4 mm, then it can be inserted under the MCAT by starting at the deepest recession. Then, the matrix is retracted laterally towards each end of the tunnel by means of mattress sutures. After positioning the matrix laterally, the site is rinsed with saline solution to remove any clot. The matrix has to be held in position using a suture (6/00).

Finally, the flap is positioned coronally to CEJ by means of suspended sutures (6/00) around the contact points.

At surgery, the duration of the full procedure will be evaluated (from anesthesia to suture).

All patients will be recall after 1, 2 and 4 weeks. They will be further recalled 3, 6 and 12 months after surgery for professional oral hygiene procedures and measurements.

ELIGIBILITY:
Inclusion Criteria:

* multiple (i.e., at least 2) Miller Class I and/or II gingival recessions located in the maxillary, with an apico-coronal extension (i.e., defect depth > 1 mm with at least one defect > 2 mm) and with at least 1 mm of residual keratinized tissue,
* good general health, with no systemic diseases that could influence the outcome of the therapy,
* healthy periodontal conditions (i.e., no presence of sites ≥ 4 mm and/or presence of intra-bony defects in the selected sites),
* adequate oral hygiene (full mouth plaque score (FMPS) of <25% at baseline (following initial oral hygiene instructions and prophylaxis),
* an adequate control of inflammation (full mouth bleeding score [FMBS]) of <25% at baseline (following initial oral hygiene instructions and prophylaxis).

Exclusion Criteria:

* subjects who currently smoke >10 cigarettes/day,
* female subjects who are nursing, pregnant, or plan to become pregnant,
* contraindication against oral surgical interventions,
* contraindication against use of Fibro-Gide (acute infection in the area of surgery and patient with collagen allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-05-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
percentage (%) of complete root coverage (CRC) | 12 months
  Ratio scale - higher values represent a better result

SECONDARY OUTCOMES:
keratinized tissue width (KTW) | 3, 6 and 12 months
  Ratio scale - higher values represent a better result
gingival thickness (GT) | 3, 6 and 12 months
  Ratio scale - higher values represent a better result
percentage of root coverage (RC %) | 3, 6 and 12 months
  Ratio scale - higher values represent a better result
post-surgical pain (PP), | 1 week after surgery
  Visual analog scale (VAS) - values from 0=[no pain] to 10=[worst pain ever]

CONTACTS AND LOCATIONS:
Overall Officials: Massimo de Sanctis, MD, Principal Investigator — Università Vita-Salute San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aroca S, Molnar B, Windisch P, Gera I, Salvi GE, Nikolidakis D, Sculean A. Treatment of multiple adjacent Miller class I and II gingival recessions with a Modified Coronally Advanced Tunnel (MCAT) technique and a collagen matrix or palatal connective tissue graft: a randomized, controlled clinical trial. J Clin Periodontol. 2013 Jul;40(7):713-20. doi: 10.1111/jcpe.12112. Epub 2013 Apr 30. PMID 23627374
- [Background] Zucchelli G, Mele M, Mazzotti C, Marzadori M, Montebugnoli L, De Sanctis M. Coronally advanced flap with and without vertical releasing incisions for the treatment of multiple gingival recessions: a comparative controlled randomized clinical trial. J Periodontol. 2009 Jul;80(7):1083-94. doi: 10.1902/jop.2009.090041. PMID 19563288
- [Background] Jepsen K, Jepsen S, Zucchelli G, Stefanini M, de Sanctis M, Baldini N, Greven B, Heinz B, Wennstrom J, Cassel B, Vignoletti F, Sanz M. Treatment of gingival recession defects with a coronally advanced flap and a xenogeneic collagen matrix: a multicenter randomized clinical trial. J Clin Periodontol. 2013 Jan;40(1):82-9. doi: 10.1111/jcpe.12019. Epub 2012 Oct 10. PMID 23050490
- [Background] Aroca S, Keglevich T, Barbieri B, Gera I, Etienne D. Clinical evaluation of a modified coronally advanced flap alone or in combination with a platelet-rich fibrin membrane for the treatment of adjacent multiple gingival recessions: a 6-month study. J Periodontol. 2009 Feb;80(2):244-52. doi: 10.1902/jop.2009.080253. PMID 19186964
- [Background] Thombre V, Koudale SB, Bhongade ML. Comparative evaluation of the effectiveness of coronally positioned flap with or without acellular dermal matrix allograft in the treatment of multiple marginal gingival recession defects. Int J Periodontics Restorative Dent. 2013 May-Jun;33(3):e88-94. doi: 10.11607/prd.1371. PMID 23593633

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT04225351/Prot_SAP_000.pdf